CLINICAL TRIAL: NCT04361695
Title: Preemptive Analgesia for Hemorrhoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2020-03-26; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Hemorrhoidectomy
MeSH Terms: interventions — Hemorrhoidectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketoprophenum (Active Comparator): A tablet with 10 mg Ketoprophenum is taken per os 2 hours before surgery
  Interventions: Procedure: Hemorrhoidectomy; Drug: Ketoprophenum
- Placebo (Placebo Comparator): A tablet containing starch is taken per os 2 hours before surgery
  Interventions: Procedure: Hemorrhoidectomy; Drug: Placebo

INTERVENTIONS:
Procedure: Hemorrhoidectomy — The patient receives spinal anaesthesia and is placed in lithotomy position. A complex of external and internal haemorrhoid or internal haemorrhoid only is excised with monopolar electrocautery or bipolar electrosurgery device. Haemorrhoid pedicle is tied with absorbable polyfilament suture. One, two or three nodes can be removed per a procedure.
Drug: Ketoprophenum — Ketoprophenum
  Arms: Ketoprophenum
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Preemptive analgesia with the spinal anesthesia allows to decrease pain in hemorrhoidectomy postoperative period. The purpose of this study is to assess the effectiveness of the use of preemptive analgesia with spinal anesthesia to decrease postoperative pain and the amount of used analgesics including opioids.

DETAILED DESCRIPTION:
Hemorrhoidectomy, as has being demonstrated to be an effective method of treatment for stage III-IV hemorrhoidal disease. However it is associated with intense postoperative pain that requires the use of multimodal analgesia. Inadequate pain control leads to the prolongation of admission, increasing the consumption of opioid analgesics, patients dissatisfaction with treatment.

According to international guidelines of pain management the target level of postoperative pain should be 3-4 or less Visual Analogue Score (VAS) points. The multimodal analgesia including Nonsteroidal Anti-Inflammatory Drugs (NSAIDs), acetaminophen and local anaesthetics are used to reach this aim.

However, there are data on effectiveness of preemptive analgesia in anorectal surgery. Preemptive analgesia allows decreasing pain in postoperative period after hemorrhoidectomy.

Ketoprophenum is used as an preemptive analgetic agent 1 hour prior to procedure.

The aim of this prospective, randomized, double-blind study is to assess the effectiveness of the use of preemptive analgesia with Ketoprophenum 10 mg 2 hours before procedure per os with spinal anaesthesia to decrease postoperative pain and the amount of used analgesics.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Patients over 18 years.
3. Symptomatic grade III-IV haemorrhoids.
4. Planned surgery: Milligan-Morgan hemorrhoidectomy

Exclusion Criteria:

1. Patient's refusal to participate in the study.
2. Pregnancy.
3. Contraindication or technical inability to perform subarachnoid anaesthesia.
4. Decompensated somatic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-02-25 (Estimated); Study Completion 2022-08-25 (Estimated)

PRIMARY OUTCOMES:
The frequency of opioid analgesics usage | 0-7 days postoperatively
  The frequency of opioid administration per day

SECONDARY OUTCOMES:
Severity of pain | 6, 12 and 24 hours after the operation, then 2 times per day up to 7th postoperative day
  The severity of the pain syndrome before defecation and after defecation reported by the patient according to Visual Analogue Score (VAS), where 0 - the minimum pain, 10 - the worst pain.
Duration of other analgesics usage | 0-7 days postoperatively
  The duration in days of systemic and topical analgesics usage
Frequency of other analgesics usage | 0-7 days postoperatively
  Times per day of systemic and topical analgesics usage
Re-admission rate | 30 days postoperatively
  The rate of patients who were re-admitted due to refractory pain
Overall quality of life | 7th and 30th days postoperatively
  Assessed with patient-reported questionnaire Short Form 36 (SF-36). A total score in each of 8 sections will be calculated and transformed into a 0-100 scale with a score of zero equivalent to maximum disability and a score of 100 equivalent to no disability
Returning to work | 30 days postoperatively
  The period of time in days from the operation to returning to work
The rate of early postoperative complications | 0-30 days postoperatively
  The rate of complications: bleeding, retention of urine, infectious complications in early postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Petr Tsarkov, Professor, Principal Investigator — Russian Society of Colorectal Surgeons
Locations (1):
- Clinic of Colorectal and Minimally Invasive Surgery, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kazachenko E, Garmanova T, Derinov A, Markaryan D, Lee H, Magbulova S, Tsarkov P. Preemptive analgesia for hemorrhoidectomy: study protocol for a prospective, randomized, double-blind trial. Trials. 2022 Jun 27;23(1):536. doi: 10.1186/s13063-022-06107-0. PMID 35761383